CLINICAL TRIAL: NCT00762463
Title: A 6-Week, Randomized, Double-Blind, Parallel-Group Study To Evaluate The Symptomatic Effects And Safety Of Celecoxib 200mg QD Compared To Diclofenac 75mg SR QD In Chinese Patients With Ankylosing Spondylitis, With 6-Week Extension Phase Treatment On Celecoxib 400 Mg QD Or Maintaining Double-Blind Phase Therapy
Brief Title: Study Of Celecoxib Or Diclofenac For Efficacy and Safety In Chinese Patients With Ankylosing Spondylitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3191348
Record Dates: First submitted 2008-09-29; First posted 2008-09-30 (Estimated); Results first posted 2011-08-23 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Celecoxib 200 mg QD (Experimental)
  Interventions: Drug: Celecoxib
- Diclofenac SR 75 mg QD (Active Comparator)
  Interventions: Drug: Diclofenac SR

INTERVENTIONS:
Drug: Celecoxib — capsule, 200 mg QD, 6-12 weeks
  Arms: Celecoxib 200 mg QD
Drug: Diclofenac SR — tablet, 75 mg QD,6-12 weeks
  Arms: Diclofenac SR 75 mg QD

SUMMARY:
This is a local, multicenter, randomized, active comparator, double-blind, parallel group study with extension will be conducted to evaluate the efficacy and safety of celecoxib versus diclofenac SR in the treatment of Chinese patients with Ankylosing Spondylitis (AS).

ELIGIBILITY:
Inclusion Criteria:

* Meet the 1984 Modified New York Criteria for Classification of Ankylosing Spondylitis
* With axial involvement
* Without peripheral joint involvement (synovitis) at the time of study entry, (excluding involvement of the hips, knees and shoulders)
* Need for daily treatment with NSAIDs during the previous 30 days before study entry

Exclusion Criteria:

* Known inflammatory enteropathy (eg, ulcerative colitis, Crohn's disease, etc)
* Presence of extra-articular manifestations (eg, uveitis, endocarditis, etc.)
* Known vertebral compression
* Need for a corset during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2009-07; Primary Completion 2010-06 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- China (4):
  - Pfizer Investigational Site, Guangzhou, Guangdong
  - Pfizer Investigational Site, Xi’an, Shanxi
  - Pfizer Investigational Site, Chengdu, Sichuan
  - Pfizer Investigational Site, Beijing

REFERENCES:
- [Derived] Huang F, Gu J, Liu Y, Zhu P, Zheng Y, Fu J, Pan S, Le S. Efficacy and safety of celecoxib in chinese patients with ankylosing spondylitis: a 6-week randomized, double-blinded study with 6-week open-label extension treatment. Curr Ther Res Clin Exp. 2014 Dec 5;76:126-33. doi: 10.1016/j.curtheres.2014.08.002. eCollection 2014 Dec. PMID 25516774
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3191348&StudyName=Study%20Of%20Celecoxib%20Or%20Diclofenac%20For%20Efficacy%20and%20Safety%20In%20Chinese%20Patients%20With%20Ankylosing%20Spondylitis

RESULTS

PARTICIPANT FLOW:
Groups:
- Celecoxib 200 mg: Celecoxib 200 milligram (mg) capsule once daily
- Diclofenac SR 75 mg: Diclofenac sustained release (SR) 75 mg tablet once daily
- Celecoxib 200 mg, Then Celecoxib 400 mg: Celecoxib 200 mg capsule once daily from baseline to Week 6 followed by Celecoxib 400 mg capsules once daily from Week 6 to Week 12
- Diclofenac SR 75 mg, Then Celecoxib 400 mg: Diclofenac SR 75 mg tablet once daily from baseline to Week 6 followed by Celecoxib 400 mg capsules once daily from Week 6 to Week 12
Period: Double-blind Phase (Baseline to Week 6)
Arm/Group | Celecoxib 200 mg | Diclofenac SR 75 mg | Celecoxib 200 mg, Then Celecoxib 400 mg | Diclofenac SR 75 mg, Then Celecoxib 400 mg
Started | 120 | 120 | 0 | 0
Completed | 113 | 110 | 0 | 0
Not Completed | 7 | 10 | 0 | 0
Not completed — Insufficient clinical response | 2 | 2 | 0 | 0
Not completed — No longer willing to participate | 3 | 4 | 0 | 0
Not completed — Adverse Event | 2 | 4 | 0 | 0
Period: Enrollment in Extension Phase (Week 6)
Arm/Group | Celecoxib 200 mg | Diclofenac SR 75 mg | Celecoxib 200 mg, Then Celecoxib 400 mg | Diclofenac SR 75 mg, Then Celecoxib 400 mg
Started | 113 | 110 | 0 | 0
Completed | 109 | 109 | 0 | 0
Not Completed | 4 | 1 | 0 | 0
Not completed — Did not sign 2nd informed consent form | 4 | 1 | 0 | 0
Period: Extension Phase (Week 6 to Week 12)
Arm/Group | Celecoxib 200 mg | Diclofenac SR 75 mg | Celecoxib 200 mg, Then Celecoxib 400 mg | Diclofenac SR 75 mg, Then Celecoxib 400 mg
Started | 55 | 55 | 54 | 54
Completed | 52 | 54 | 50 | 52
Not Completed | 3 | 1 | 4 | 2
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0
Not completed — Insufficient clinical response | 1 | 1 | 0 | 1
Not completed — No longer willing to participate | 1 | 0 | 3 | 0
Not completed — Other | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Celecoxib 200 mg: Celecoxib 200 mg capsule once daily
- Diclofenac SR 75 mg: Diclofenac SR 75 mg tablet once daily
- Total: Total of all reporting groups
Arm/Group | Celecoxib 200 mg | Diclofenac SR 75 mg | Total
Number analyzed (Participants) | 120 | 120 | 240
Age, Customized [Number; unit: participants]
  18 - 44 years | 109 | 109 | 218
  45 - 64 years | 11 | 11 | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 19 | 34
  Male | 105 | 101 | 206

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Participant's Assessment of Global Pain Intensity at Week 6
Description: 100-millimeter (mm) Visual Analog Scale (VAS) score specified participant's assessment of overall pain intensity in the previous 48 hours, in response to the following question "What has been your global pain intensity in the last 48 hours?" 0=no pain to 100=worst pain. Change from baseline of less than (<) 0 indicated improvement.
Time Frame: Baseline, Week 6
Population: Per-Protocol (PP): All randomized participants who received at least one dose of study medication, and had global pain intensity assessment at Week 6 and no major protocol deviations.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Celecoxib 200 mg | Diclofenac SR 75 mg
Number analyzed (Participants) | 111 | 108
mm | -23.8 (1.98) | -27.1 (2.02)
Statistical Analysis 1: Comparison: Celecoxib 200 mg vs Diclofenac SR 75 mg; Null hypothesis: Least Squares (LS) mean difference between Celecoxib 200 mg once daily versus Diclofenac SR 75 mg once daily on change in Global Pain Intensity from baseline to Week 6 was at least 10 mm. Corresponding alternative hypothesis: This difference was <10 mm. For the non-inferiority test, power was 80% and significance level was 0.025 (1-sided); Test type: Non-Inferiority or Equivalence — LS mean difference calculated as LS mean change for Celecoxib 200 mg once daily minus LS mean change for Diclofenac SR 75 mg once daily. Non-inferiority was declared if the upper bound of the 95% confidence interval was <10 mm; p = 0.0085, ANCOVA; Analysis of covariance (ANCOVA); factors: treatment group and study center; covariate: baseline Patient's Assessment of Global Pain Intensity score; LS Mean Difference = 3.3, 95% CI 2-sided [-2.2 to 8.8], Standard Error of Mean 2.79

2. Primary Outcome: Participant's Assessment of Global Pain Intensity at Baseline
Description: 100-mm VAS scores specified participant's assessment of global pain intensity in the previous 48 hours, in response to the following question "What has been your global pain intensity in the last 48 hours?" 0=no pain to 100=worst pain. Lower scores indicated less pain.
Time Frame: Baseline
Population: PP
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Celecoxib 200 mg | Diclofenac SR 75 mg
Number analyzed (Participants) | 111 | 108
mm | 62.9 (12.68) | 63.6 (13.38)

3. Secondary Outcome: Change From Baseline in Participant's Assessment of Global Pain Intensity at Weeks 2 and 4
Description: 100-mm VAS score specified participant's assessment of overall pain intensity in the previous 48 hours, in response to the following question "What has been your global pain intensity in the last 48 hours?" 0=no pain to 100=worst pain. Change from baseline of <0 indicated improvement.
Time Frame: Baseline, Weeks 2, 4
Population: Full Analysis Set (FAS). Number of participants analyzed (N) = total evaluable participants. n = evaluable participants at that time point.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Celecoxib 200 mg | Diclofenac SR 75 mg
Number analyzed (Participants) | 117 | 115
mm
  Week 2 (n=116, 115) | -18.6 (1.78) | -17.9 (1.79)
  Week 4 (n=117, 115) | -20.7 (1.86) | -23.3 (1.89)
Statistical Analysis 1: Comparison: Celecoxib 200 mg vs Diclofenac SR 75 mg; Change from baseline to Week 2. The p-value is for the null hypothesis test H0: u1=u2 vs. H1: u1 is not equal to u2; Test type: Superiority or Other; p = 0.7849, ANCOVA; Change from baseline analyzed using ANCOVA with treatment group and investigational centers as factors and baseline value as a covariate; LS Mean Difference = -0.7, 95% CI 2-sided [-5.6 to 4.2], Standard Error of Mean 2.50
Statistical Analysis 2: Comparison: Celecoxib 200 mg vs Diclofenac SR 75 mg; Change from baseline to Week 4. The p-value is for the null hypothesis test H0: u1=u2 vs. H1: u1 is not equal to u2; Test type: Superiority or Other; p = 0.3223, ANCOVA; Change from baseline was analyzed using ANCOVA with treatment group and investigational centers as factors and baseline value as a covariate; LS Mean Difference = 2.6, 95% CI 2-sided [-2.6 to 7.8], Standard Error of Mean 2.62

4. Secondary Outcome: Change From Baseline in Participant's Assessment of Global Pain Intensity at Week 12
Description: 100-mm VAS score specified participant's assessment of overall pain intensity in the previous 48 hours, in response to the following question "What has been your global pain intensity in the last 48 hours?" 0=no pain to 100=worst pain. Lower scores indicated less pain. Change from baseline of <0 indicated improvement.
Time Frame: Baseline, Week 12
Population: FAS. n = evaluable participants at that time point.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Celecoxib 200 mg | Diclofenac SR 75 mg | Celecoxib 200 mg, Then Celecoxib 400 mg | Diclofenac SR 75 mg, Then Celecoxib 400 mg
Number analyzed (Participants) | 55 | 55 | 54 | 54
mm
  Baseline (n=55, 55, 54, 54) | 63.4 (13.58) | 61.1 (13.08) | 63.4 (12.05) | 65.6 (13.26)
  Change from Baseline at Week 12 (n=52, 54, 46, 51) | -28.4 (21.39) | -30.9 (24.24) | -20.8 (21.86) | -28.1 (25.96)

5. Secondary Outcome: Change From Baseline in Participant's Global Assessment of Disease Activity at Weeks 2, 4, and 6
Description: 5-point Likert scale scores specified participant's current situation in response to the following question "Considering all the ways your Ankylosing Spondylitis affects you, how are you doing today?" 1=very good to 5=very poor. Change from baseline <0 indicated improvement.
Time Frame: Baseline, Weeks 2, 4, 6
Population: FAS. N = total evaluable participants. n = evaluable participants at that time point.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Celecoxib 200 mg | Diclofenac SR 75 mg
Number analyzed (Participants) | 117 | 115
units on a scale
  Week 2 (n=116, 115) | -0.4 (0.06) | -0.4 (0.06)
  Week 4 (n=117, 115) | -0.3 (0.06) | -0.4 (0.06)
  Week 6 (n=117, 115) | -0.3 (0.06) | -0.4 (0.06)
Statistical Analysis 1: Comparison: Celecoxib 200 mg vs Diclofenac SR 75 mg; Change from baseline to Week 2. The p-value is for the null hypothesis test H0: u1=u2 vs. H1: u1 is not equal to u2; Test type: Superiority or Other; p = 0.8938, ANCOVA; [statistical method as in outcome 3, analysis 2]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.15 to 0.17], Standard Error of Mean 0.08
Statistical Analysis 2: Comparison: Celecoxib 200 mg vs Diclofenac SR 75 mg; Change from baseline to Week 4. The p-value is for the null hypothesis test H0: u1=u2 vs. H1: u1 is not equal to u2; Test type: Superiority or Other; p = 0.0426, ANCOVA; [statistical method as in outcome 3, analysis 2]; LS Mean Difference = 0.2, 95% CI 2-sided [0.01 to 0.31], Standard Error of Mean 0.08
Statistical Analysis 3: Comparison: Celecoxib 200 mg vs Diclofenac SR 75 mg; Change from baseline to Week 6. The p-value is for the null hypothesis test H0: u1=u2 vs. H1: u1 is not equal to u2; Test type: Superiority or Other; p = 0.1502, ANCOVA; [statistical method as in outcome 3, analysis 2]; LS Mean Difference = 0.1, 95% CI 2-sided [-0.05 to 0.29], Standard Error of Mean 0.09

6. Secondary Outcome: Change From Baseline in Participant's Global Assessment of Disease Activity at Week 12
Description: 5-point Likert scale scores specified participant's current situation in response to the following question "Considering all the ways your Ankylosing Spondylitis affects you, how are you doing today?" 1=very good to 5=very poor. Lower scores indicated better health. Change from baseline <0 indicated improvement.
Time Frame: Baseline, Week 12
Population: FAS. n = evaluable participants at that time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Celecoxib 200 mg | Diclofenac SR 75 mg | Celecoxib 200 mg, Then Celecoxib 400 mg | Diclofenac SR 75 mg, Then Celecoxib 400 mg
Number analyzed (Participants) | 55 | 55 | 54 | 54
units on a scale
  Baseline (n=55, 55, 54, 54) | 3.1 (0.83) | 3.0 (0.64) | 3.2 (0.66) | 3.2 (0.70)
  Change from Baseline at Week 12 (n=52, 54, 46, 51) | -0.6 (0.99) | -0.6 (0.78) | -0.4 (0.71) | -0.6 (0.96)

7. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Disease Activity at Weeks 2, 4, and 6
Description: 5-point Likert scale scores specified physician's subjective assessment on how overall ankylosing spondylitis appeared at the time of participant's visit and participant's disease signs. 1=very good to 5=very poor. Change from baseline <0 indicated improvement.
Time Frame: Baseline, Weeks 2, 4, 6
Population: FAS. N = total evaluable participants. n = evaluable participants at that time point.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Celecoxib 200 mg | Diclofenac SR 75 mg
Number analyzed (Participants) | 117 | 115
units on a scale
  Week 2 (n=116, 115) | -0.4 (0.05) | -0.4 (0.05)
  Week 4 (n=117, 115) | -0.4 (0.05) | -0.5 (0.05)
  Week 6 (n=117, 115) | -0.5 (0.06) | -0.5 (0.06)
Statistical Analysis 1: Comparison: Celecoxib 200 mg vs Diclofenac SR 75 mg; Change from baseline to Week 2. The p-value is for the null hypothesis test H0: u1=u2 vs. H1: u1 is not equal to u2; Test type: Superiority or Other; p = 0.5945, ANCOVA; [statistical method as in outcome 3, analysis 2]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.2 to 0.1], Standard Error of Mean 0.07
Statistical Analysis 2: Comparison: Celecoxib 200 mg vs Diclofenac SR 75 mg; Change from baseline to Week 4. The p-value is for the null hypothesis test H0: u1=u2 vs. H1: u1 is not equal to u2; Test type: Superiority or Other; p = 0.3427, ANCOVA; [statistical method as in outcome 3, analysis 2]; LS Mean Difference = 0.1, 95% CI 2-sided [-0.1 to 0.2], Standard Error of Mean 0.07
Statistical Analysis 3: Comparison: Celecoxib 200 mg vs Diclofenac SR 75 mg; Change from baseline to Week 6. The p-value is for the null hypothesis test H0: u1=u2 vs. H1: u1 is not equal to u2; Test type: Superiority or Other; p = 0.6522, ANCOVA; [statistical method as in outcome 3, analysis 2]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.1 to 0.2], Standard Error of Mean 0.08

8. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Disease Activity at Week 12
Description: 5-point Likert scale scores specified physician's subjective assessment on how the overall ankylosing spondylitis appeared at the time of the participant's visit and participant's disease signs. 1=very good to 5=very poor. Lower scores indicated better health. Change from baseline <0 indicated improvement.
Time Frame: Baseline, Week 12
Population: FAS. n = evaluable participants at that time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Celecoxib 200 mg | Diclofenac SR 75 mg | Celecoxib 200 mg, Then Celecoxib 400 mg | Diclofenac SR 75 mg, Then Celecoxib 400 mg
Number analyzed (Participants) | 55 | 55 | 54 | 54
units on a scale
  Baseline (n=55, 55, 54, 54) | 3.2 (0.57) | 3.0 (0.45) | 3.2 (0.43) | 3.3 (0.50)
  Change from Baseline at Week 12 (n=52, 54, 46, 51) | -0.7 (0.60) | -0.5 (0.64) | -0.5 (0.51) | -0.7 (0.75)

9. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Functional Index (BASFI) at Weeks 2, 4, and 6
Description: Bath Ankylosing Spondylitis Functional Index (BASFI) was comprised of 10 specific questions, each answered on a 10-mm VAS scale. 0=easy to 10=impossible. BASFI score was defined as the mean of the scaled responses to these 10 questions. Change from baseline <0 indicated improvement.
Time Frame: Baseline, Weeks 2, 4, 6
Population: FAS. N = total evaluable participants. n = evaluable participants at that time point.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Celecoxib 200 mg | Diclofenac SR 75 mg
Number analyzed (Participants) | 117 | 115
mm
  Week 2 (n=116, 115) | -0.3 (0.13) | -0.3 (0.13)
  Week 4 (n=117, 115) | -0.4 (0.14) | -0.6 (0.14)
  Week 6 (n=117, 115) | -0.5 (0.15) | -0.8 (0.15)
Statistical Analysis 1: Comparison: Celecoxib 200 mg vs Diclofenac SR 75 mg; Change from baseline to Week 2. The p-value is for the null hypothesis test H0: u1=u2 vs. H1: u1 is not equal to u2; Test type: Superiority or Other; p = 0.9358, ANCOVA; [statistical method as in outcome 3, analysis 2]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.3 to 0.4], Standard Error of Mean 0.18
Statistical Analysis 2: Comparison: Celecoxib 200 mg vs Diclofenac SR 75 mg; Change from baseline to Week 4. The p-value is for the null hypothesis test H0: u1=u2 vs. H1: u1 is not equal to u2; Test type: Superiority or Other; p = 0.5916, ANCOVA; [statistical method as in outcome 3, analysis 2]; LS Mean Difference = 0.1, 95% CI 2-sided [-0.3 to 0.5], Standard Error of Mean 0.20
Statistical Analysis 3: Comparison: Celecoxib 200 mg vs Diclofenac SR 75 mg; Change from baseline to Week 6. The p-value is for the null hypothesis test H0: u1=u2 vs. H1: u1 is not equal to u2; Test type: Superiority or Other; p = 0.1790, ANCOVA; [statistical method as in outcome 3, analysis 2]; LS Mean Difference = 0.3, 95% CI 2-sided [-0.1 to 0.7], Standard Error of Mean 0.20

10. Secondary Outcome: Change From Baseline in BASFI at Week 12
Description: BASFI was comprised of 10 specific questions, each answered on a 10-mm VAS scale. 0=easy to 10=impossible. BASFI score was defined as the mean of the scaled responses to these 10 questions. Lower scores indicated better functional health. Change from baseline <0 indicated improvement.
Time Frame: Baseline, Week 12
Population: FAS. n = evaluable participants at that time point.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Celecoxib 200 mg | Diclofenac SR 75 mg | Celecoxib 200 mg, Then Celecoxib 400 mg | Diclofenac SR 75 mg, Then Celecoxib 400 mg
Number analyzed (Participants) | 55 | 55 | 54 | 54
mm
  Baseline (n=55, 55, 54, 54) | 3.4 (1.98) | 3.5 (2.13) | 3.5 (1.83) | 3.5 (2.25)
  Change from Baseline at Week 12 (n=52, 54, 46, 51) | -0.9 (1.78) | -1.0 (1.64) | -0.6 (1.97) | -1.0 (2.30)

11. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) at Weeks 2, 4, and 6
Description: Baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) was comprised of 6 specific questions, each answered on a 10-mm VAS scale. Scores for the first 5 questions: 0=none to 10=severe. Score for the sixth question: 0=0 hours to 10=2 hours. BASDAI score was defined as the mean of the scaled responses to these 6 questions. Change from baseline <0 indicated improvement.
Time Frame: Baseline, Weeks 2, 4, 6
Population: FAS. N = total evaluable participants. n = evaluable participants at that time point.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Celecoxib 200 mg | Diclofenac SR 75 mg
Number analyzed (Participants) | 117 | 115
mm
  Week 2 (n=116, 115) | -0.8 (0.14) | -0.9 (0.14)
  Week 4 (n=117, 115) | -0.9 (0.15) | -1.1 (0.15)
  Week 6 (n=117, 115) | -1.1 (0.16) | -1.4 (0.16)
Statistical Analysis 1: Comparison: Celecoxib 200 mg vs Diclofenac SR 75 mg; Change from baseline to Week 2. The p-value is for the null hypothesis test H0: u1=u2 vs. H1: u1 is not equal to u2; Test type: Superiority or Other; p = 0.6335, ANCOVA; [statistical method as in outcome 3, analysis 2]; LS Mean Difference = 0.1, 95% CI 2-sided [-0.3 to 0.5], Standard Error of Mean 0.20
Statistical Analysis 2: Comparison: Celecoxib 200 mg vs Diclofenac SR 75 mg; Change from baseline to Week 4. The p-value is for the null hypothesis test H0: u1=u2 vs. H1: u1 is not equal to u2; Test type: Superiority or Other; p = 0.2729, ANCOVA; [statistical method as in outcome 3, analysis 2]; LS Mean Difference = 0.2, 95% CI 2-sided [-0.2 to 0.6], Standard Error of Mean 0.21
Statistical Analysis 3: Comparison: Celecoxib 200 mg vs Diclofenac SR 75 mg; Change from baseline to Week 6. The p-value is for the null hypothesis test H0: u1=u2 vs. H1: u1 is not equal to u2; Test type: Superiority or Other; p = 0.1559, ANCOVA; [statistical method as in outcome 3, analysis 2]; LS Mean Difference = 0.3, 95% CI 2-sided [-0.1 to 0.8], Standard Error of Mean 0.22

12. Secondary Outcome: Change From Baseline in BASDAI at Week 12
Description: BASDAI is comprised of 6 specific questions, each answered on a 10-mm VAS. Scores for the first 5 questions: 0=none to 10=severe. Score for the sixth question: 0=0 hours to 10=2 hours. BASDAI score was defined as the mean of the scaled responses to these 6 questions. Lower scores indicated better health. Change from baseline <0 indicated improvement.
Time Frame: Baseline, Week 12
Population: FAS. n = evaluable participants at that time point.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Celecoxib 200 mg | Diclofenac SR 75 mg | Celecoxib 200 mg, Then Celecoxib 400 mg | Diclofenac SR 75 mg, Then Celecoxib 400 mg
Number analyzed (Participants) | 55 | 55 | 54 | 54
mm
  Baseline (n=55, 55, 54, 54) | 4.71 (1.79) | 4.9 (1.80) | 4.7 (1.48) | 4.9 (1.88)
  Change from Baseline at Week 12 (n=52, 54, 46, 51) | -1.7 (1.86) | -2.1 (1.94) | -0.6 (1.87) | -1.4 (2.14)

13. Secondary Outcome: Percentages of Participants Responding to Assessment in Ankylosing Spondylitis (ASAS)-20
Description: Percentages of participants who demonstrated an improvement of greater than or equal to (≥) 20% from baseline and an absolute improvement of ≥10 mm from baseline on a 100-mm VAS in ≥3 of the 4 domains proposed by the Ankylosing Spondylitis Assessment Working Group (ASAS-20).
Time Frame: Weeks 2, 4, 6, 12
Population: FAS. N = total evaluable participants. n = evaluable participants at that time point.
Measure: Number; unit: percentage of participants
Groups:
- Diclofenac 75 mg, Then Celecoxib 400 mg: Diclofenac SR 75 mg tablet once daily from baseline to Week 6 and Celecoxib 400 mg once daily from Week 6 to Week 12
Arm/Group | Celecoxib 200 mg | Diclofenac SR 75 mg | Celecoxib 200 mg, Then Celecoxib 400 mg | Diclofenac 75 mg, Then Celecoxib 400 mg
Number analyzed (Participants) | 116 | 114 | 55 | 55
percentage of participants
  Week 2 (n=115, 114) | 23.5 | 25.4 | 0 | 0
  Week 4 (n=116, 114) | 26.7 | 31.6 | 0 | 0
  Week 6 (n=54, 54, 54, 54) | 40.7 | 42.6 | 22.2 | 29.6
  Week 12 (n=51, 53, 46, 51) | 49.0 | 47.2 | 32.6 | 37.3

14. Secondary Outcome: Change From Baseline in Nocturnal Pain at Weeks 2, 4, and 6
Description: 100-mm VAS scores specified participant's nocturnal pain in response to the following question "Did you have any pain in the neck, back or hips during the previous night?" 0=no pain to 100=worst pain possible. Change from baseline <0 indicated improvement.
Time Frame: Baseline, Weeks 2, 4, 6
Population: FAS. N = total evaluable participants. n = evaluable participants at that time point.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Celecoxib 200 mg | Diclofenac SR 75 mg
Number analyzed (Participants) | 117 | 115
mm
  Week 2 (n=116, 115) | -12.0 (1.90) | -16.3 (1.91)
  Week 4 (n=117, 115) | -14.5 (1.94) | -17.1 (1.96)
  Week 6 (n=117, 115) | -15.4 (1.95) | -19.4 (1.98)
Statistical Analysis 1: Comparison: Celecoxib 200 mg vs Diclofenac SR 75 mg; Change from baseline to Week 2. The p-value is for the null hypothesis test H0: u1=u2 vs. H1: u1 is not equal to u2; Test type: Superiority or Other; p = 0.1111, ANCOVA; [statistical method as in outcome 3, analysis 2]; LS Mean Difference = 4.3, 95% CI 2-sided [-1.0 to 9.5], Standard Error of Mean 2.67
Statistical Analysis 2: Comparison: Celecoxib 200 mg vs Diclofenac SR 75 mg; Change from baseline to Week 4. The p-value is for the null hypothesis test H0: u1=u2 vs. H1: u1 is not equal to u2; Test type: Superiority or Other; p = 0.3574, ANCOVA; [statistical method as in outcome 3, analysis 2]; LS Mean Difference = 2.5, 95% CI 2-sided [-2.9 to 7.9], Standard Error of Mean 2.74
Statistical Analysis 3: Comparison: Celecoxib 200 mg vs Diclofenac SR 75 mg; Change from baseline to Week 6. The p-value is for the null hypothesis test H0: u1=u2 vs. H1: u1 is not equal to u2; Test type: Superiority or Other; p = 0.1464, ANCOVA; [statistical method as in outcome 3, analysis 2]; LS Mean Difference = 4.0, 95% CI 2-sided [-1.4 to 9.5], Standard Error of Mean 2.76

15. Secondary Outcome: Change From Baseline in Nocturnal Pain at Week 12
Description: 100-mm VAS scores specified participant's nocturnal pain in response to the following question "Did you have any pain in the neck, back or hips during the previous night?" 0=no pain to 100=worst pain possible. Lower scores indicated less pain. Change from baseline <0 indicated improvement.
Time Frame: Baseline, Week 12
Population: FAS. n = evaluable participants at that time point.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Celecoxib 200 mg | Diclofenac SR 75 mg | Celecoxib 200 mg, Then Celecoxib 400 mg | Diclofenac SR 75 mg, Then Celecoxib 400 mg
Number analyzed (Participants) | 55 | 55 | 54 | 54
mm
  Baseline (n=55, 55, 54, 54) | 52.2 (20.45) | 55.1 (19.24) | 54.5 (20.14) | 61.5 (19.17)
  Change from Baseline at Week 12 (n=52, 54, 46, 51) | -19.4 (22.54) | -27.5 (25.62) | -12.5 (20.31) | -22.6 (30.36)

16. Secondary Outcome: Change From Baseline in Fingertips to Floor Distance at Weeks 2, 4, and 6
Description: Fingertips to floor distance measured in centimeter (cm) from the tip of the fingers to the floor with participants standing erect and feet together, knees as straight as possible, then bending forward as far as possible with fingers reaching towards the floor. The better of 2 tries was recorded. Change from baseline <0 indicated improvement.
Time Frame: Baseline, Weeks 2, 4, 6
Population: FAS. N = total evaluable participants. n = evaluable participants at that time point.
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | Celecoxib 200 mg | Diclofenac SR 75 mg
Number analyzed (Participants) | 118 | 115
cm
  Week 2 (n=117, 115) | -1.6 (0.62) | -1.6 (0.62)
  Week 4 (n=118, 115) | -1.9 (0.69) | -2.2 (0.71)
  Week 6 (n=118, 115) | -2.8 (0.67) | -3.1 (0.69)
Statistical Analysis 1: Comparison: Celecoxib 200 mg vs Diclofenac SR 75 mg; Change from baseline to Week 2. The p-value is for the null hypothesis test H0: u1=u2 vs. H1: u1 is not equal to u2; Test type: Superiority or Other; p = 0.9641, ANCOVA; [statistical method as in outcome 3, analysis 2]; LS Mean Difference = 0.0, 95% CI 2-sided [-1.7 to 1.8], Standard Error of Mean 0.87
Statistical Analysis 2: Comparison: Celecoxib 200 mg vs Diclofenac SR 75 mg; Change from baseline to Week 4. The p-value is for the null hypothesis test H0: u1=u2 vs. H1: u1 is not equal to u2; Test type: Superiority or Other; p = 0.7749, ANCOVA; [statistical method as in outcome 3, analysis 2]; LS Mean Difference = 0.3, 95% CI 2-sided [-1.6 to 2.2], Standard Error of Mean 0.98
Statistical Analysis 3: Comparison: Celecoxib 200 mg vs Diclofenac SR 75 mg; Change from baseline to Week 6. The p-value is for the null hypothesis test H0: u1=u2 vs. H1: u1 is not equal to u2; Test type: Superiority or Other; p = 0.7529, ANCOVA; [statistical method as in outcome 3, analysis 2]; LS Mean Difference = 0.3, 95% CI 2-sided [-1.6 to 2.2], Standard Error of Mean 0.95

17. Secondary Outcome: Change From Baseline in Fingertips to Floor Distance at Week 12
Description: Fingertips to floor distance measured in cm from the tip of the fingers to the floor with participant standing erect and feet together, knees as straight as possible, then bending forward as far as possible with fingers reaching towards the floor. The better of 2 tries was recorded. Lower scores indicated better health. Change from baseline <0 represented improvement.
Time Frame: Baseline, Week 12
Population: FAS. n = evaluable participants at that time point.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Celecoxib 200 mg | Diclofenac SR 75 mg | Celecoxib 200 mg, Then Celecoxib 400 mg | Diclofenac SR 75 mg, Then Celecoxib 400 mg
Number analyzed (Participants) | 55 | 55 | 54 | 54
cm
  Baseline (n=55, 55, 54, 54) | 14.8 (12.89) | 17.6 (15.23) | 22.9 (19.49) | 14.6 (14.48)
  Change from Baseline at Week 12 (n=52, 54, 46, 51) | -3.0 (9.38) | -3.7 (6.82) | -3.1 (8.18) | -1.3 (7.75)

18. Secondary Outcome: Change From Baseline in Chest Expansion at Weeks 2, 4, and 6
Description: Chest expansion, measured in cm, is defined as the difference in thoracic circumference during full expiration versus full inspiration, measured at the fourth intercostal space (nipple line). The better of 2 tries was recorded. Change from baseline greater than (>) 0 represented improvement.
Time Frame: Baseline, Weeks 2, 4, 6
Population: FAS. N = total evaluable participants. n = evaluable participants at that time point.
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | Celecoxib 200 mg | Diclofenac SR 75 mg
Number analyzed (Participants) | 118 | 115
cm
  Week 2 (n=117, 115) | 0.2 (0.08) | 0.3 (0.08)
  Week 4 (n=118, 115) | 0.6 (0.09) | 0.4 (0.09)
  Week 6 (n=118, 115) | 0.7 (0.10) | 0.6 (0.10)
Statistical Analysis 1: Comparison: Celecoxib 200 mg vs Diclofenac SR 75 mg; Change from baseline to Week 2. The p-value is for the null hypothesis test H0: u1=u2 vs. H1: u1 is not equal to u2; Test type: Superiority or Other; p = 0.8780, ANCOVA; [statistical method as in outcome 3, analysis 2]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.2 to 0.2], Standard Error of Mean 0.11
Statistical Analysis 2: Comparison: Celecoxib 200 mg vs Diclofenac SR 75 mg; Change from baseline to Week 4. The p-value is for the null hypothesis test H0: u1=u2 vs. H1: u1 is not equal to u2; Test type: Superiority or Other; p = 0.2202, ANCOVA; [statistical method as in outcome 3, analysis 2]; LS Mean Difference = 0.2, 95% CI 2-sided [-0.1 to 0.4], Standard Error of Mean 0.13
Statistical Analysis 3: Comparison: Celecoxib 200 mg vs Diclofenac SR 75 mg; Change from baseline to Week 6. The p-value is for the null hypothesis test H0: u1=u2 vs. H1: u1 is not equal to u2; Test type: Superiority or Other; p = 0.5340, ANCOVA; [statistical method as in outcome 3, analysis 2]; LS Mean Difference = 0.1, 95% CI 2-sided [-0.2 to 0.4], Standard Error of Mean 0.14

19. Secondary Outcome: Change From Baseline in Chest Expansion at Week 12
Description: Chest expansion, measured in cm, is defined as the difference in thoracic circumference during full expiration versus full inspiration, measured at the fourth intercostal space (nipple line). The better of 2 tries was recorded. Higher scores indicate better health. Change from baseline greater than (>) 0 represented improvement.
Time Frame: Baseline, Week 12
Population: FAS. n = evaluable participants at that time point.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Celecoxib 200 mg | Diclofenac SR 75 mg | Celecoxib 200 mg, Then Celecoxib 400 mg | Diclofenac SR 75 mg, Then Celecoxib 400 mg
Number analyzed (Participants) | 55 | 55 | 54 | 54
cm
  Baseline (n=55, 55, 54, 54) | 3.9 (1.93) | 3.8 (1.63) | 3.6 (1.82) | 3.8 (1.62)
  Change from Baseline at Week 12 (n=52, 54, 46, 51) | 0.8 (1.26) | 0.8 (1.39) | 0.8 (1.29) | 0.8 (1.02)

20. Secondary Outcome: Change From Baseline in Erythrocyte Sedimentation Rate (ESR) at Week 6
Description: Erythrocyte Sedimentation Rate (ESR) was a laboratory test that providee a non-specific measure of inflammation. The test assessed the rate at which red blood cells fell in a test tube and was measured in millimeter per hour (mm/h). Change from baseline <0 indicated improvement.
Time Frame: Baseline, Week 6
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: mm/h
Arm/Group | Celecoxib 200 mg | Diclofenac SR 75 mg
Number analyzed (Participants) | 108 | 110
mm/h | -2.5 (1.30) | -1.8 (1.30)
Statistical Analysis 1: Comparison: Celecoxib 200 mg vs Diclofenac SR 75 mg; The p-value is for the null hypothesis test H0: u1=u2 vs. H1: u1 is not equal to u2; Test type: Superiority or Other; p = 0.7003, ANCOVA; [statistical method as in outcome 3, analysis 1]; LS Mean Difference = -0.7, 95% CI 2-sided [-4.3 to 2.9], Standard Error of Mean 1.81

21. Secondary Outcome: Change From Baseline in ESR at Week 12
Description: ESR was a laboratory test that provided a non-specific measure of inflammation. The test assessed the rate at which red blood cells fell in a test tube. Lower values indicated better health. Change from baseline <0 indicated improvement.
Time Frame: Baseline, Week 12
Population: FAS. n = evaluable participants at that time point.
Measure: Mean (Standard Deviation); unit: mm/h
Arm/Group | Celecoxib 200 mg | Diclofenac SR 75 mg | Celecoxib 200 mg, Then Celecoxib 400 mg | Diclofenac SR 75 mg, Then Celecoxib 400 mg
Number analyzed (Participants) | 54 | 54 | 52 | 54
mm/h
  Baseline (n=54, 54, 52, 54) | 20.9 (14.60) | 20.8 (18.98) | 22.8 (21.99) | 23.6 (19.64)
  Change from Baseline at Week 12 (n=45, 44, 41, 43) | -3.5 (13.96) | -1.3 (11.14) | -6.3 (13.46) | -0.7 (19.47)

22. Secondary Outcome: Change From Baseline in C-Reactive Protein (CRP) at Week 6
Description: C-Reactive Protein (CRP) was a marker of inflammation, measured in milligram per liter (mg/L). Change from baseline <0 indicated improvement.
Time Frame: Baseline, 6 Weeks
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: mg/L
Arm/Group | Celecoxib 200 mg | Diclofenac SR 75 mg
Number analyzed (Participants) | 109 | 110
mg/L | -4.16 (1.587) | -2.72 (1.600)
Statistical Analysis 1: Comparison: Celecoxib 200 mg vs Diclofenac SR 75 mg; The p-value is for the null hypothesis test H0: u1=u2 vs. H1: u1 is not equal to u2; Test type: Superiority or Other; p = 0.5183, ANCOVA; [statistical method as in outcome 3, analysis 1]; LS Mean Difference = -1.44, 95% CI 2-sided [-5.82 to 2.94], Standard Error of Mean 2.221

23. Secondary Outcome: Change From Baseline in CRP at Week 12
Description: CRP was a marker of inflammation. Lower values indicated better health. Change from baseline <0 indicated improvement.
Time Frame: Baseline, Week 12
Population: FAS. n = evaluable participants at that time point.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Celecoxib 200 mg | Diclofenac SR 75 mg | Celecoxib 200 mg, Then Celecoxib 400 mg | Diclofenac SR 75 mg, Then Celecoxib 400 mg
Number analyzed (Participants) | 53 | 55 | 53 | 54
mg/L
  Baseline (n=53, 55, 53, 54) | 18.53 (28.749) | 15.84 (20.464) | 18.80 (25.774) | 21.01 (21.360)
  Change from Baseline at Week 12 (n=47, 49, 42, 47) | -4.58 (9.682) | -2.99 (13.242) | -4.77 (24.656) | -2.13 (20.879)

24. Secondary Outcome: Percentage of Participants With Concomitant Use of Paracetamol
Description: Percentage of participants who concomitantly took at least 1 paracetamol tablet as rescue medication at Week 6
Time Frame: Week 6
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Celecoxib 200 mg | Diclofenac SR 75 mg
Number analyzed (Participants) | 120 | 120
percentage of participants | 2.5 | 0.0

25. Secondary Outcome: Percentage of Days With Concomitant Administration of Paracetamol
Description: Calculated as days on rescue medication divided by days of exposure in the study at the end of Week 6.
Time Frame: Week 6
Population: FAS
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Celecoxib 200 mg | Diclofenac SR 75 mg
Number analyzed (Participants) | 120 | 120
percentage of days | 0.1 (0.08) | 0.0 (0.00)

26. Secondary Outcome: Paracetamol Tablets Taken Per Day by Participant
Description: Calculated as the total number of paracetamol tablets taken divided by days of exposure in the study.
Time Frame: Week 6
Population: FAS
Measure: Mean (Standard Deviation); unit: tablets per day
Arm/Group | Celecoxib 200 mg | Diclofenac SR 75 mg
Number analyzed (Participants) | 120 | 120
tablets per day | 0.2 (0.16) | 0.0 (0.00)

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious AE (SAE). However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Groups:
- Celecoxib 200 mg: Celecoxib 200 mg capsule once daily from baseline to Week 6
- Diclofenac SR 75 mg: Diclofenac SR 75 mg tablet once daily from baseline to Week 6
- Celecoxib 200 mg, Then Celecoxib 200 mg: Celecoxib 200 mg capsule once daily from baseline to Week 6, followed by Celecoxib 200 mg capsule once daily from Week 6 to Week 12
- Diclofenac SR 75 mg, Then Diclofenac SR 75 mg: Diclofenac SR 75 mg tablet once daily from baseline to Week 6 followed by Diclofenac SR 75 mg tablet once daily from Week 6 to Week 12
- Celecoxib 200 mg, Then Celecoxib 400 mg: Celecoxib 200 mg capsule once daily from baseline to Week 6, followed by Celecoxib 400 mg capsules once daily from Week 6 to Week 12
- Diclofenac SR 75 mg, Then Celecoxib 400 mg: Diclofenac SR 75 mg tablet once daily from baseline to Week 6, followed by Celecoxib 400 mg capsules once daily from Week 6 to Week 12
Arm/Group | Celecoxib 200 mg | Diclofenac SR 75 mg | Celecoxib 200 mg, Then Celecoxib 200 mg | Diclofenac SR 75 mg, Then Diclofenac SR 75 mg | Celecoxib 200 mg, Then Celecoxib 400 mg | Diclofenac SR 75 mg, Then Celecoxib 400 mg
Serious Adverse Events (participants affected / at risk) | 0/120 | 0/120 | 0/54 | 0/55 | 0/53 | 0/54
Other Adverse Events (participants affected / at risk) | 11/120 | 9/120 | 0/54 | 6/55 | 5/53 | 6/54
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Celecoxib 200 mg (N=120) | Diclofenac SR 75 mg (N=120) | Celecoxib 200 mg, Then Celecoxib 200 mg (N=54) | Diclofenac SR 75 mg, Then Diclofenac SR 75 mg (N=55) | Celecoxib 200 mg, Then Celecoxib 400 mg (N=53) | Diclofenac SR 75 mg, Then Celecoxib 400 mg (N=54)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Wolff-Parkinson-White Syndrome (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Uveitis (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 2 | 0 | 1 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 1 | 0 | 0 | 0 | 2
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 2 | 1 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Red blood cell urine positive (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
VIIth nerve paralysis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The protocol does not specify time points for secondary endpoints; these are described in the statistical analysis plan.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.